CLINICAL TRIAL: NCT01133301
Title: Naltrexone in the Treatment of Dissociative Symptoms in Patients With Borderline Personality Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: University of Freiburg (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Naltrexone-BPD; nal-diss-bpd (Other: Intern)
Record Dates: First submitted 2010-05-17; First posted 2010-05-28 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2010-05

CONDITIONS: Borderline Personality Disorder; Dissociation
Keywords: Borderline Personality Disorder; Dissociation; Naltrexone
MeSH Terms: conditions — Borderline Personality Disorder; Dissociative Disorders | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naltrexone-Placebo (Active Comparator): In the first three weeks of the study, 50 mg Naltrexone will be administrated, the following three three weeks placebo will be administrated.
  Interventions: Drug: Naltrexone; Drug: Placebo
- Placebo-Naltrexone (Placebo Comparator): The first three weeks, placebo will be administrated, the following three weeks 50 mg Naltrexone will be administrated.
  Interventions: Drug: Naltrexone; Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — 50 mg/d Naltrexone will be administrated during three weeks.
Drug: Placebo — During 3 weeks of the study, Placebo will be administrated (daily)

SUMMARY:
Our study aims at contributing to a valid appraisal of the magnitude of naltrexone efficacy as an antidissociative agent by using a double-blind randomized controlled trial.

DETAILED DESCRIPTION:
Patients were randomized into two groups starting with either 3 weeks of 50 mg/d naltrexone or with 3 weeks of placebo. In either case the active treatment phases (weeks 1-6) were followed by one week of placebo. The major purpose of weeks 1-2 and 4-5, respectively, was to achieve a steady state during the active treatment. The primary comparisons of psychopathology under naltrexone and placebo refer to the weeks following the intended achievement of a steady state (weeks 3 and 6, respectively).

6 weeks of treatment were split into two phases: (A) 3 weeks of pharmacologically active treatment with naltrexone and (B) 3 weeks of pharmacologically inactive treatment with placebo (cross-over design). The sequence of the two treatment phases was randomized and concealed from both the patients and the health care professionals. In both cases, the last week ("Week 7") was without pharmacological intervention.

The primary outcome was based on the DSS, a reliable and valid self-rating instrument to assess dissociative experiences and inner tension during the last 24 hours (Stiglmayr et al. 2001) Mean scores for intensity (ranging from 0="no" to 9="very strong") and for duration (average time during which a particular symptom was present during the last 24 hours (in %)) were calculated for (a) dissociation (calculated from 21 Likert type items) and of (b) aversive inner tension (one item).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of BPD according to DSM-IV
* DES score ≥ 18
* Female gender
* Age between 18 and 50 years

Exclusion Criteria:

* Lifetime diagnosis of schizophrenia, psychotic or delusional disorder
* Current major depressive episode
* Lifetime diagnosis opioid dependence
* Current diagnosis opioid abuse
* Liver insufficiency or hepatitis
* Other major medical or neurological medical condition
* Pregnancy or lactation
* Psychotropic medication within two weeks before and during the trial (fluoxetine 4 weeks, lithium 8 weeks)
* Concomitant treatment with opioid analgetics
* Hypersensitivity to naltrexone

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 1998-08; Primary Completion 2001-08 (Actual); Study Completion 2001-10 (Actual)

PRIMARY OUTCOMES:
Dissociation Tension Scale (DSS), a reliable and valid self-rating instrument to assess dissociative experiences and inner tension during the last 24 hours (Stiglmayr et al. 2001) | Oct. 1998-Oct 2001

SECONDARY OUTCOMES:
The number, the method, and the severity of non-suicidal self-injurious acts during the last week.
  The number, method and the severity of non-suicidal self-injurious acts are documented at the end of each week.
Number and intensity of flashbacks during the last week.
  The number and intensity of flashbacks are documented at the end of each week

CONTACTS AND LOCATIONS:
Overall Officials: Christian Schmahl, MD, Study Chair — Central Institute of Mental Health, Dep. of Psychosomatic and Psychotherapeutic Medicine
Locations (1):
- Department of Psychiatry and Psychotherapy, University of Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Stoffers-Winterling JM, Storebo OJ, Pereira Ribeiro J, Kongerslev MT, Vollm BA, Mattivi JT, Faltinsen E, Todorovac A, Jorgensen MS, Callesen HE, Sales CP, Schaug JP, Simonsen E, Lieb K. Pharmacological interventions for people with borderline personality disorder. Cochrane Database Syst Rev. 2022 Nov 14;11(11):CD012956. doi: 10.1002/14651858.CD012956.pub2. PMID 36375174